CLINICAL TRIAL: NCT01863953
Title: A Safety and Efficacy Study of Fixed-Combination Bimatoprost and Brimonidine in Chronic Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-082
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate; Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed-Combination Bimatoprost/Brimonidine (Experimental): One drop fixed-combination bimatoprost/brimonidine in each eye twice daily for 6 weeks.
  Interventions: Drug: Fixed-Combination Bimatoprost/Brimonidine
- Bimatoprost Ophthalmic Solution 0.01% and Vehicle (Active Comparator): One drop bimatoprost ophthalmic solution 0.01% in each eye in the evening and vehicle ophthalmic solution in each eye in the morning daily for 6 weeks.
  Interventions: Drug: Bimatoprost Ophthalmic Solution 0.01%; Drug: Vehicle Ophthalmic Solution
- Brimonidine Tartrate Ophthalmic Solution 0.2% (Active Comparator): One drop brimonidine tartrate ophthalmic solution 0.2% in each eye twice daily for 6 weeks.
  Interventions: Drug: Brimonidine Tartrate Ophthalmic Solution 0.2%

INTERVENTIONS:
Drug: Fixed-Combination Bimatoprost/Brimonidine — One drop fixed-combination bimatoprost/brimonidine in each eye twice daily for 6 weeks.
  Arms: Fixed-Combination Bimatoprost/Brimonidine
Drug: Bimatoprost Ophthalmic Solution 0.01% — One drop bimatoprost ophthalmic solution 0.01% in each eye in the evening for 6 weeks.
  Other Names: LUMIGAN
  Arms: Bimatoprost Ophthalmic Solution 0.01% and Vehicle
Drug: Vehicle Ophthalmic Solution — One drop vehicle ophthalmic solution in each eye in the morning daily for 6 weeks.
  Arms: Bimatoprost Ophthalmic Solution 0.01% and Vehicle
Drug: Brimonidine Tartrate Ophthalmic Solution 0.2% — One drop brimonidine tartrate ophthalmic solution 0.2% in each eye twice daily for 6 weeks.
  Other Names: ALPHAGAN
  Arms: Brimonidine Tartrate Ophthalmic Solution 0.2%

SUMMARY:
This is a safety and efficacy study of fixed-combination bimatoprost and brimonidine compared with LUMIGAN® and ALPHAGAN® in patients with chronic glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension or glaucoma
* Requires intraocular pressure (IOP)-lowering therapy

Exclusion Criteria:

* Cataract surgery in one eye
* Ocular laser or intraocular surgery within 6 months
* Refractive surgery in either eye
* Anticipated use of contact lenses during the study
* Expected use of artificial tears during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2%
Started | 38 | 36 | 38
Completed | 38 | 36 | 37
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2% | Total
Number analyzed (Participants) | 38 | 36 | 38 | 112
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 0 | 0 | 1
  Between 45 and 65 years | 21 | 14 | 20 | 55
  >65 years | 16 | 22 | 18 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 25 | 67
  Male | 18 | 14 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Eye Mean Diurnal Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. Average eye mean diurnal IOP is the mean of the average eye IOPs (average IOP of the right and left eyes) at hours 0, 2, 4, 8 and 12. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase in IOP (worsening).
Time Frame: Baseline, Day 42
Population: Modified Intent to Treat: all randomized and treated patients who had baseline and at least 1 postbaseline IOP assessment
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2%
Number analyzed (Participants) | 38 | 36 | 38
Millimeters of Mercury (mmHg)
  Baseline | 24.54 (1.712) | 24.38 (2.022) | 24.29 (1.457)
  Change from Baseline at Day 42 (N=38, 36, 37) | -6.79 (2.277) | -6.63 (2.284) | -3.92 (2.574)

2. Secondary Outcome: Change From Baseline in Average Eye Mean Diurnal IOP
Description: as for outcome 1
Time Frame: Baseline, Day 14, Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2%
Number analyzed (Participants) | 38 | 36 | 38
mmHg
  Baseline | 24.54 (1.712) | 24.38 (2.022) | 24.29 (1.457)
  Change from Baseline at Day 14 | -7.63 (2.152) | -6.79 (1.997) | -4.67 (2.944)
  Change from Baseline at Day 28 | -7.25 (2.328) | -6.98 (2.260) | -4.22 (2.869)

3. Secondary Outcome: Average Eye Mean Diurnal IOP
Description: IOP is a measurement of the fluid pressure inside the eye. Average eye mean diurnal IOP is the mean of the average eye IOPs (average IOP of the right and left eyes) at hours 0, 2, 4, 8 and 12.
Time Frame: Day 14, Day 28, Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2%
Number analyzed (Participants) | 38 | 36 | 38
mmHg
  Day 14 | 16.91 (2.004) | 17.59 (2.363) | 19.61 (2.572)
  Day 28 | 17.29 (2.588) | 17.40 (2.549) | 20.06 (2.540)
  Day 42 (N=38, 36, 37) | 17.75 (2.505) | 17.76 (2.467) | 20.34 (2.218)

ADVERSE EVENTS:
Description: Treatment emergent adverse events (TEAE) are reported and include all adverse events (AEs) and serious adverse events (SAEs) that began or worsened after study treatment.
Arm/Group | Fixed-Combination Bimatoprost/Brimonidine | Bimatoprost Ophthalmic Solution 0.01% and Vehicle | Brimonidine Tartrate Ophthalmic Solution 0.2%
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/36 | 1/38
Other Adverse Events (participants affected / at risk) | 27/38 | 25/36 | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed-Combination Bimatoprost/Brimonidine (N=38) | Bimatoprost Ophthalmic Solution 0.01% and Vehicle (N=36) | Brimonidine Tartrate Ophthalmic Solution 0.2% (N=38)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed-Combination Bimatoprost/Brimonidine (N=38) | Bimatoprost Ophthalmic Solution 0.01% and Vehicle (N=36) | Brimonidine Tartrate Ophthalmic Solution 0.2% (N=38)
Conjunctival Hyperaemia (Eye disorders) | 18 | 16 | 2
Eye Pruritus (Eye disorders) | 5 | 5 | 3
Eye Discharge (Eye disorders) | 3 | 1 | 1
Blepharospasm (Eye disorders) | 3 | 0 | 0
Punctate Keratitis (Eye disorders) | 2 | 4 | 2
Eye Pain (Eye disorders) | 2 | 1 | 2
Instillation Site Pruritus (General disorders) | 2 | 1 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 2 | 0 | 1
Instillation Site Lacrimation (General disorders) | 2 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 2
Eye Irritation (Eye disorders) | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 4
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.